CLINICAL TRIAL: NCT03964272
Title: A Feasibility Study on the Safety and Preliminary Efficacy of Bilateral Subthalamotomy Using the ExAblate Transcranial System to Treat the Cardinal Motor Features of Parkinson's Disease
Brief Title: A Feasibility Study on the Safety and Preliminary Efficacy of Bilateral Subthalamotomy Using MRgFUS for Treatment of PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PD010B
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Neurologic Manifestations
Keywords: MRgFUS; ExAblate; Parkinsons Disease; Sub-Thalamotomy
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExAblate 4000 System (Experimental): Exablate bilateral treatment for Parkinson's Disease Motor Features
  Interventions: Device: Exablate Bilateral Subthalamotomy

INTERVENTIONS:
Device: Exablate Bilateral Subthalamotomy — Exablate bilateral treatment for Parkinson's Disease Motor Features
  Other Names: MRgFUS; Subthalamotomy

SUMMARY:
The objective of this study is to test the safety and preliminary efficacy of staged bilateral subthalamotomy performed using the ExAblate Transcranial System for the treatment of Parkinson's disease (PD) motor features

DETAILED DESCRIPTION:
The objective of this study is to evaluate the incidence and severity of adverse events (AE/AEs) associated with ExAblate Transcranial Magnetic Resonance Guided Focused Ultrasound (MRgFUS) bilateral staged subthalamotomy for the treatment of PD motor features. To determine the effectiveness of the ExAblate Transcranial staged bilateral subthalamotomy to treat cardinal motor features of subjects with PD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 30 years or older
2. Able and willing to give consent and able to attend all study visits
3. A confirmed diagnosis of Parkinsons Disease
4. Subjects that have received unilateral subthalamotomy at least 6 month before the inclusion in bilateral subthalamotomy and present parkinsonian symptoms
5. Able to localize subthalamic nucleus on MRI for treatment
6. Able to communicate sensations during the ExAblate MRgFUS procedure

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 2.5 or greater
2. Presence of severe dyskinesia as noted by MDS-UPDRS scores
3. Presence of other central neurodegenerative disease
4. Parkinsonian symptoms are a side effect from neuroleptic medications
5. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse
6. History of a bleeding disorder or receiving anticoagulant
7. Subjects with advanced kidney disease or on dialysis
8. Subjects with known intolerance or allergies to the MRI contrast agents.
9. Presence of unknown or MRI unsafe devices anywhere in the body.
10. History of multiple strokes, or a stroke within past 6 months
11. Subjects with a history of seizures within the past year
12. Subjects with malignant brain tumors
13. Women who are pregnant or nursing

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Events | Treatment through 6 month
  To evaluate the incidence and severity of adverse events (AE/AEs) associated with ExAblate subthalamotomy for the treatment of PD motor features.
Primary Efficacy: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Off Medication Status | Treatment through 6 month
  Effectiveness of the ExAblate Transcranial staged bilateral subthalamotomy by analyzing mean change (reduction from baseline to 6 months) in the motor MDS-UPDRS score in the treated group as compared with baseline in the off-medication condition

SECONDARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) On Medication Status | Treatment through 6 month
  - Mean change (reduction) in the motor MDS-UPDRS score in the on-medication condition (when applicable)
MDS-UPDRS | Treatment through 12 month
  - Mean change (reduction) in specific PD motor features (i.e., tremor, rigidity and akinesia according to MDS-UPDRS III subscores)
MDS-UPDRS (Part I, II and IV) | Treatment through 6 month
  MDS UPDRS I, II and IV
Quality of life assessment | Treatment through 6 month
  Improved Quality of life assessment with the PDQ39

CONTACTS AND LOCATIONS:
Overall Officials: Raul Martinez, MD, Principal Investigator — CINAC-Hospital HM Puerta del Sur
Locations (1):
- Hospital Universitario HM Puerta Del Sur. CINAC, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No